CLINICAL TRIAL: NCT06852768
Title: A Double-Masked, Randomized, Placebo-Controlled Study of the Safety, Tolerability, and Efficacy of d-MAPPS™ Ophthalmic Solution in the Treatment of Chronic Ocular Graft-Versus-Host Disease (oGVHD)
Brief Title: Study of d-MAPPS™ Ophthalmic Solution, Safety, Tolerability, and Efficacy in the Treatment of Chronic Ocular Graft-Versus-Host Disease (oGVHD)
Acronym: oGVHD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regenerative Ocular Immunobiologics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30066
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: oGHVD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- This arm randomizes the actual drug to the patient. (Active Comparator): Based on randomization, d-MAPPS™ will be self-administered, 2 drops into each eye four times (QID) a day for ninety (90) days.
  Interventions: Biological: d-MAPPS
- This arm randomizes the placebo to the patient. (Placebo Comparator): Based on randomization Placebo/sterile water, will be self-administered, 2 drops into each eye four times (QID) a day for ninety (90) days.
  Interventions: Biological: Placebo
- Both patient and PI are masked. (Other): Upon acceptance into the study, the sponsor will be notified, and the patient will be randomized to the treatment or placebo arm. Randomization Code Key will have limited access to only authorized personnel. Based on the results of the randomization selection, the sponsor will provide the appropriate subject number and lot coded eyedropper bottles containing d-MAPPS™ or Placebo/sterile water to the doctor for dissemination.
  Interventions: Biological: d-MAPPS; Biological: Placebo; Other: PI and Patient Masked

INTERVENTIONS:
Biological: d-MAPPS — Based on randomization d-MAPPS, will be self-administered, 2 drops into each eye four times a day (QID) a day for ninety (90) days.
  Arms: Both patient and PI are masked.; This arm randomizes the actual drug to the patient.
Biological: Placebo — Based on randomization, Placebo, will be self-administered, 2 drops into each eye four times (QID) a day for ninety (90) days.
  Arms: Both patient and PI are masked.; This arm randomizes the placebo to the patient.
Other: PI and Patient Masked — Both the PI and the participant are masked on the drug administered.
  Arms: Both patient and PI are masked.

SUMMARY:
A Double-Masked, Randomized, Placebo-Controlled Study of the Safety, Tolerability, and Efficacy of d-MAPPS™ Ophthalmic Solution in the Treatment of Chronic Ocular Graft-Versus-Host Disease (oGHVD)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with study assessments for the full duration of the study.
* Patients may be using bilateral scleral lenses and/or bilateral punctal plugs at the time of accrual.
* Minimum Oxford Schema grad of ≥ 1 in at least one eye.
* OSDI scored of ≥ 22.
* UNC DEMS score of ≥ 3.
* In good stable overall health.

Exclusion Criteria:

* History of Rheumatoid Arthritis, Lupus, Scleroderma.
* Ocular or periocular malignancy.
* Significant change, as judged by the principal investigator, in systemic immunosuppressive regimen within 2 weeks of study entry.
* Any history of topical tacrolimus use.
* Any change in dosage of tetracycline compounds (tetracycline, doxycycline, and minocycline) within the last month.
* Any change in frequency of preserved anti-glaucoma medications within 2 weeks of study entry.
* Current use of topical steroids more than twice a day.
* Corneal epithelial defect > 1mm2.
* Any history of herpetic keratitis.
* Participation in another simultaneous medical research study.
* Signs of current infection, including fever and current treatment with antibiotics.
* All vaccination including COVID are prohibited during this study.
* Signs of current infection, including fever and current treatment with antibiotics.
* All vaccinations including COVID are prohibited during this study.
* Intra-ocular surgery or ocular laser surgery within 3 months.
* Women who are pregnant, breastfeeding, or plan to become pregnant while participating in the study. If of childbearing potential, unwillingness to use effective birth control while participating in the study.
* Any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline utilizing University of North Carolina Dry Eye Management Scale (UNC DEMS) Scores | Through study completion, an average of 4 months.
  The UNC Dry Eye Management Scale (DEMS) helps evaluate different aspects of DED, including symptoms, severity, and impact on daily life. Dry eye symptoms such as grittiness, dryness, foreign body sensation, redness, tearing, and irritation. The UNC DEMS is used in clinical settings to inform treatment decisions and monitor the effectiveness of interventions. UNC DEMS scores are on a scale from 1-10, with 10 being the most severe. The changes will be evaluated from baseline and at timepoints 30 ±5 days, 60 ±5 days and 90 ±5 days.
Changes from Baseline utilizing Ocular Surface Disease Index (OSDI) | Through study completion, an average of 4 months.
  Ocular Surface Disease Index (OSDI) Questionnaire is a 12-question survey used to measure the symptoms of dry eye disease. Each of the 12 individual questions rate each of the dry eye symptoms on a 0-4 scale. The results are calculated in an overall scale that ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms. The changes will be evaluated from baseline and at timepoints 30 ±5 days, 60 ±5 days and 90 ±5 days.

SECONDARY OUTCOMES:
Changes from baseline utilizing the NIH Eye Score for chronic oGVHD | Through study completion, an average of 4 months.
  The NIH Eye Score is a recommended measure, as it detects improvement or worsening in ocular chronic GVHD. Scoring from 0 to 3 is based on symptoms, need for eye drops, and use of therapeutic procedures or devices.
Changes from Baseline Oxford Schema for Corneal and Conjunctival Stain Grades | Through study completion, an average of 4 months.
  Oxford Schema for Corneal and Conjunctival Staining is a diagnostic test that looks for signs of damage or dryness in the eye. It involves a doctor applying dye to the eye to show areas of damage on its surface. The Oxford grading scale divides corneal staining into 6 groups according to severity: 0 = absent, I = minimal, II = mild, III = moderate, IV = marked, and V = severe. The changes will be evaluated from baseline and at timepoints 30 ±5 days, 60 ±5 days and 90±5 days.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Beverly Hills Institute of Ophthalmology, Beverly Hills, California
  - Beach Eye Medical Group, Huntington Beach, California
  - Regenerative Ocular Immunobiologics, LLC., Palm Harbor, Florida
  - Glenn Eye Center, Lexington, Kentucky
  - Eyewell, LLC., Boston, Massachusetts